CLINICAL TRIAL: NCT04481633
Title: Real-life Evaluation of the Efficacy of Pre-exposure Treatment With Hydroxy-Chloroquine on the Risk and Severity of COVID-19 Infection in Patients Receiving Long-term Treatment for Systemic Lupus Erythematosus and/or Gougerot's Disease
Brief Title: Efficacy of Pre-exposure Treatment With Hydroxy-Chloroquine on the Risk and Severity of COVID-19 Infection
Acronym: PREPCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/20/0186; 2020-A01906-33 (Other: N° ID-RCB)
Record Dates: First submitted 2020-07-21; First posted 2020-07-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
Keywords: lupus erythematous disease; prophylaxis; pre-emptive therapy; Hydroxy-Chloroquine
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient treated with Hydroxy-chloroquine (Other): patients treated with Hydroxy-Chloroquine (HC) with or without immunosuppressants (IS)(HC+ group, n=400)
  Interventions: Diagnostic Test: COVID 19 serology; Other: COVID 19 Self-Questionnaire
- Patient without treatment with Hydroxy-chloroquine (Other): patients without treatment with Hydroxy-Chloroquine with or without immunosuppressants
  Interventions: Diagnostic Test: COVID 19 serology; Other: COVID 19 Self-Questionnaire

INTERVENTIONS:
Diagnostic Test: COVID 19 serology — Diagnosis of Covid-19 past infection will be made by serology
Other: COVID 19 Self-Questionnaire — COVID 19 Self-Questionnaire

SUMMARY:
There is a pandemic in the world by COVID-19. Currently, the pharmacological curative or prophylactic treatments for this infection are not known. Recent studies have suggested that Hydroxy-Chloroquine could be effective in vitro and in vivo against COVID-19. The main objective of this study is to assess in patients with autoimmune disease treated with long course Hydroxy-Chloroquine initiated before the pandemic COVID-19 had an independent protective effect on the risk or the severity of infection with COVID-19.

DETAILED DESCRIPTION:
A pre- or post-exposure treatment strategy has been validated in some infectious diseases. In particular, in HIV infection, this type of prophylactic treatment reduces the rate of infection in at-risk populations. The first studies from Chinese show that in case of immunosuppression or immunosuppressive treatment, whatever the causal pathology, COVID-19 infection is more severe. The present study presents a population of patients with lupus (SLE) or Gougerot's disease (SGD) who are treated for a long time, with Hydroxy-Chloroquine. The protective effect against COVID-19 infection of Hydroxy-Chloroquine compared to populations not exposed to this drug requires to be assessed in patients and their control groups under or without immunosuppressive treatments.

It is hypothesized that long-term treatment with Hydroxy-Chloroquine in SLE or SGD taken in its usual indication before the onset of the pandemic could decrease the number of COVID19 infections and/or the intensity of the disease.

ELIGIBILITY:
Inclusion Criteria:

Group with hydroxychloroquine treatment (HC +):

* LED/SG diagnosed
* Treatment with Hydroxy-Chloroquine in the 3 months before and during the outbreak at COVID 19, at least in December 2019. Patients may have treatment with immunosuppressants in combination with Hydroxy-Chloroquine.
* COVID19 diagnostic questionnaire and available serology result.

Group without hydroxychloroquine treatment (HC-) :

* No Hydroxy-Chloroquine intake for more than 12 months

  --> HC- without an immunosuppressant
* Viral hepatitis C cured for more than 12 months or primitive bile cholangitis (CBP) whose diagnosis is based on international criteria.
* Non-significant liver fibrosis assessed either by historical histology or by fibroscan with non-significant liver fibrosis Metavir - F3 (at last available examination)
* No Hydroxy-Chloroquine, or immunosuppressants have been taken for more than 12 months.
* COVID19 diagnostic questionnaire and COVID19 serology result available.

  -->HC- with an immunosuppressant
* Diagnosis of LED/SG according to the CAB criteria revised in 1997 or autoimmune hepatitis according to the international criteria validated in 2008.
* Patients treated with immunosuppressants for at least three months before the start of the pandemic at COVID 19, at least since December 2019.
* COVID19 diagnostic questionnaire and available serology result.

Exclusion Criteria:

* Anti-CD20 or Cyclophosphamide taken during the six months prior to the completion of the COVID 19 serology.
* Refusal of a blood test for antibodies to COVID-19.
* Protected adults
* Pregnant or breastfeeding women.
* Lack of health insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Rate of patients with positive anti-COVID19 serology | Day 1
  Rate of patients with positive anti-COVID19 serology with or without Hydroxy-Chloroquine.

SECONDARY OUTCOMES:
Rate of patients with symptomatic or severe (hospitalization) form of infection | Day 1
  Rate of patients with symptomatic or severe (hospitalization) form of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent ALRIC, Pr, Principal Investigator — University Hospital, Toulouse
Locations (12):
- France (12):
  - Limoges university Hospital, Limoges
  - Montpellier University Hospital, Montpellier
  - Pitié Salpêtrière Hospital - Hépatologie, Paris
  - Pitié Salpêtrière Hospital - Médecine interne, Paris
  - Haut-Lévêque Hospital - Gastro-entérologie, Pessac
  - Haut-Lévêque Hospital - Médecine interne, Pessac
  - Joseph Ducuing Hospital - Médecine interne, Toulouse
  - Toulouse university Hospital - Larrey Dermatologie, Toulouse
  - Toulouse University Hospital - Rhumatologie, Toulouse
  - Toulouse University Hospital, Toulouse
  - University Hospital of Toulouse - Rangueil Médecine interne, Toulouse
  - University hospital Toulouse - Purpan Médecine interne, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Result] Alric L, Brusq C, Migueres M, Faure S, Lebray P, Viallard JF, Chauveau D, Sailler L, Berard E, Pugnet G, Cacoub P; Prepcov study. Evaluation of the effects of pre-exposure treatment with hydroxychloroquine on the risk of COVID-19 infection and on the efficacy of anti-COVID-19 vaccination during lupus or Gougerot-Sjogren's disease: Prepcov multicentre trial. Lupus Sci Med. 2025 Mar 5;12(1):e001435. doi: 10.1136/lupus-2024-001435. PMID 40044500